CLINICAL TRIAL: NCT01461772
Title: Comparison of Concurrent Chemoradiation Therapy With Weekly Cisplatin and Concurrent Chemoradiation Therapy With Weekly Carboplatin in Locally Advanced Cervical Cancer: Phase III Multicenter Prospective Randomized Controlled Trial
Brief Title: Efficacy and Safety Study of Concurrent Chemoradiation Therapy to Treat Locally Advanced Cervical Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Because of very slow rate of enrollement
Sponsor: Asan Medical Center (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Joo-Hyun Nam, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCRTCICA-CXCA
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy; Carboplatin; Cisplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CCRT weekly carboplatin (Experimental): Concurrent chemoradiation therapy with weekly carboplatin
  Interventions: Radiation: Radiation therapy; Drug: Carboplatin
- CCRT weekly cisplatin (Active Comparator): Concurrent chemoradiation therapy with weekly cisplatin
  Interventions: Radiation: Radiation therapy; Drug: Cisplatin

INTERVENTIONS:
Radiation: Radiation therapy — pelvic radiation therapy (Extended filed radiation therapy and addition of brachytherapy is allowed)
Drug: Carboplatin — carboplatin 130mg/m2BSA on day 1,8,15,22,29,and 36
  Arms: CCRT weekly carboplatin
Drug: Cisplatin — Cisplatin 40mg/m2BSA on day 1,8,15,22,29,and 36
  Arms: CCRT weekly cisplatin

SUMMARY:
Concurrent chemoradiation therapy with weekly cisplatin is the current standard treatment for patients with locally advanced cervical cancer. However, weekly cisplatin is related to renal toxicity and not convenient regimen. Recently, carboplatin has proved to be a good radiosensitizer and less renal toxicity. Weekly carboplatin is more convenient regimen for both patients and physicians. Weekly carboplatin may have similar efficacy with weekly cisplatin and may have more favorable toxicity profile. Therefore, the investigators aimed to evaluate the efficacy and safety of concurrent chemoradiation with weekly carboplatin in patients with locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histologically confirmed cervical cancer
* One of following histologic types Squamous carcinoma, adenocarcinoma, adenosquamous carcinoma
* Age: 20-75 years
* GOG performance status: 0-2
* Adequate organ function Bone marrow: WBC ≥ 3,000/mm3, ANC ≥ 1,500/mm3, Platelet ≥ 100X103/mm3, Hb ≥ 10.0 g/dl Kidney: Creatinine < 1.25 × UNL, Liver : AST, ALT < 3 × UNL, T- bilirubin < 1.5 mg/ mm3
* Contraception during study treatment
* Informed consent

Exclusion Criteria:

* Previous chemotherapy or pelvic radiation therapy
* Hormone therapy within 4 weeks
* Concomitant malignancy within 5 years except cured basal cell carcinoma of skin
* Uncontrolled medical disease
* Pregnant or lactating woman
* Etc.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Response rate | 3 months after completion of study treatment

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | Before each chemotherapy, an average of 1 week
Disease-free survival | 2 years after completion of study treatment
Overall survival | 2 years after completion of study treatment
Quality of life | 3 months after completion of study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea